CLINICAL TRIAL: NCT06910384
Title: An Open Label Study of STR04 in Participants With Amyotrophic Lateral Sclerosis
Brief Title: A Study of STRO4 in Patients Amyotrophic Lateral Sclerosis (ALS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: organizational restructure
Sponsor: New England Cell Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NECT 24-03
Record Dates: First submitted 2025-03-07; First posted 2025-04-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm, Open Label (Other)
  Interventions: Biological: STR04

INTERVENTIONS:
Biological: STR04 — autologous bone-marrow-derived mesenchymal stem cells

SUMMARY:
This study intends to evaluate the safety and efficacy of STR04 administered intravenously in participants with Amyotrophic Lateral Sclerosis.

DETAILED DESCRIPTION:
This study is a 69 week open label study of autologous bone-marrow-derived mesenchymal stem cells (STR04) in participants with ALS.

Participants will undergo a screening visit, followed by collection of peripheral blood and bone marrow for the manufacture of STR04. Once manufacturing is successfully completed, participants will have a Baseline visit followed by 4 doses of STR04, one dose every 12 weeks. Participants will have a final assessments 12 weeks after the 4th dose.

ELIGIBILITY:
Inclusion:

* "Definite" or "Probable" ALS according to the Revised El Escorial criteria (Airlie House)
* ALS severity grade 1 or 2 according to the Japan ALS severity classification.
* ALSFRS-R scores of 2 or more for all items, with scores of 4 for all breathing- related items (i.e., dyspnea, orthopnea, respiratory insufficiency).
* Within 2 years of ALS onset.
* %FVC of 80% or more.
* Aged 18 to ≤75 years at the time of informed consent.

Exclusion:

* Current Viral Infection (e.g. HBV, HCV, HIV, HTLV-1, HPVB19, syphilis, COVID- 19).
* Current low blood cell counts
* History of cancer, congenital malformations, or chromosomal abnormalities
* History of allergy to penicillin or streptomycin, or other serious allergies.
* Current poor medical condition, due to endocrine disease, metabolic disease, immune disease, blood disease, psychiatric disorders, neurological diseases, cardiovascular diseases, respiratory diseases, gastrointestinal diseases, musculoskeletal or connective tissue diseases, renal or urogenital diseases.
* History of intracranial lesions, or stenosis, dissection or severe atherosclerotic disease of a blood vessel in the head or neck.
* Current uncontrolled hypertension.
* Prior treatment with a cell or gene therapy.
* Currently participating in any other clinical trial.
* Women who are pregnant, breastfeeding, or plan to become pregnant during study participation
* Men with plan for their partner to become pregnant during study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-08-12 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Change in Amyotrophic Lateral Sclerosis Functional Rating Scale Score | 25 weeks

SECONDARY OUTCOMES:
Change in Amyotrophic Lateral Sclerosis Functional Rating Scale Score | 49 weeks
Change in Percent-predicted forced vital capacity (%FVC) | From Baseline to 25 weeks and 49 weeks
Change in Manual Muscle Test (MMT) | From Baseline to 25 weeks and 49 weeks
Change in Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40) | From Baseline to 25 weeks and 49 weeks
Change in plasma neurofilament light (NfL) | From Baseline to 25 weeks and 49 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alan Jacobs, MD, PhD, Study Director — New England Cell Therapeutics, Inc.
Locations (1):
- National Neuromuscular Research Institute, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No